CLINICAL TRIAL: NCT00736333
Title: Observational Program of Caelyx in MBC - Prevention and Treatment of PPE and Infusion Reactions
Brief Title: A Study to Evaluate Safety and Tolerability in Patients With Metastatic Breast Cancer Receiving Treatment With Caelyx (Study P04878)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04878
Record Dates: First submitted 2008-07-25; First posted 2008-08-15 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pegylated Liposomal Doxorubicin: Subjects with metastatic breast cancer
  Interventions: Drug: Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — Pegylated Liposomal Doxorubicin (Caelyx) 50 mg/m^2, given for up to 6 cycles
  Other Names: SCH 200746

SUMMARY:
This is a study to evaluate the safety and tolerability of Caelyx used for the treatment of metastatic breast cancer (MBC), focusing on infusion reaction and palmar-plantar erythrodysesthesia (PPE).

DETAILED DESCRIPTION:
Patients selected by investigator according to clinical routine

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer

Exclusion Criteria:

* History of hypersensitivity to Caelyx or its components
* Women who are pregnant or breast-feeding
* Patients with severe myelosuppression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegylated Liposomal Doxorubicin: Pegylated liposomal doxorubicin 50 mg/m^2 given every 4 weeks for up to 6 cycles
Period: Overall Study
Arm/Group | Pegylated Liposomal Doxorubicin
Started | 167
Completed | 56
Not Completed | 111
Not completed — Did Not Receive Drug or Not Documented | 7
Not completed — Data Missing | 2
Not completed — Tumor Progression | 75
Not completed — Toxicity | 6
Not completed — Withdrawal by Subject | 10
Not completed — Death | 7
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated for the intent-to-treat (ITT) population only (those who received at least one dose of study medication).
  years | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender information was available only for the ITT population.
  Participants
    Female | 159
    Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infusion Reactions (IR)
Description: Infusion reaction was defined as an allergic reaction or anaphylactoid reaction characterized by shortness of breath, hypotension, back pain, chest pain, chills, flush, sweating, fever, nausea, dizziness, rash, pruritis, or tachycardia.
Time Frame: Day 1 up to Week 24
Population: Safety population (those who received at least one dose of study medication)
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Participants | 7

2. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: CR and PR were documented according to the clinical standards of each site.
Time Frame: Day 1 up to 24 weeks
Population: Intent-to-treat (those who received at least one dose of study medication)
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Participants
  CR | 2
  PR | 29

3. Primary Outcome: Percent of Participants Taking Premedication for Prevention of IR
Description: Premedications for prevention of IR included corticosteroids, serotonin-3 receptor antagonists (anti-emetics), histamine-1 receptor blockers, and histamine-2 receptor blockers.
Time Frame: Day 1, immediately prior to receiving first dose of pegylated liposomal doxorubicin
Population: Safety population (those who received at least one dose of study medication)
Measure: Number; unit: Percent of participants
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Percent of participants
  Corticosteroids | 96.3
  Serotonin-3 receptor antagonists (anti-emetics) | 97.5
  Histamine-1 receptor blockers | 15.6
  Histamine-2 receptor blockers | 36.3

4. Primary Outcome: Number of Participants With Pre-existing Allergic Conditions Who Experienced an IR
Description: Allergic conditions included food allergies, drug allergies, allergic rhinitis, histamine allergy, neurodermatitis, and chronic idiopathic urticaria.
Time Frame: Cycles 1 & 3 (Week 4 & Week 12)
Population: Safety population (those who received at least one dose of study medication)
Measure: Number; unit: Participants
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Participants | 0

5. Primary Outcome: Number of Occurrences of Palmar-plantar Erythrodysesthesia (PPE)
Description: PPE was defined as a dermatological adverse event characterized by swelling, pain, edema, erythema, desquamation, that may have ultimately resulted in fissuring and ulceration, involving fingers, toes, palms, plantar aspects of the feet, and other pressure-sensitive areas of the skin.
Time Frame: Up to 24 weeks
Population: Safety population (those who received at least one dose of study medication)
Measure: Number; unit: Occurrences
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Occurrences | 91

6. Primary Outcome: Number of Times Premedications Were Given for Prevention of PPE
Description: Pre-medications given included oral dexamethasone, vitamin B6, and other not clearly defined medications.
Time Frame: Day 1 up to 24 weeks
Population: Safety population (those who received at least one dose of study medication)
Measure: Number; unit: Number of times premedication was given
Arm/Group | Pegylated Liposomal Doxorubicin
Number analyzed (Participants) | 160
Number of times premedication was given
  Oral dexamethasone | 66
  Vitamin B6 | 70
  Other | 49

ADVERSE EVENTS:
Description: The safety data were from the safety population (those who received at least one dose of study medication).
Arm/Group | Pegylated Liposomal Doxorubicin
Serious Adverse Events (participants affected / at risk) | 5/160
Other Adverse Events (participants affected / at risk) | 9/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Liposomal Doxorubicin (N=160)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
General physical health deterioration (General disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Liposomal Doxorubicin (N=160)
Stomatitis (Gastrointestinal disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No